CLINICAL TRIAL: NCT06393790
Title: Health Effects of a Strength Training Protocol in Women With Fibromyalgia and Healthy Individuals.
Brief Title: Strength Training Protocol in Fibromyalgia Women
Acronym: FM PROTOCOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of Murcia (Other)
Collaborators: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Carmen Daniela Quero Calero, PhD, Catholic University of Murcia
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TC/03-23; TC/03-23 (Registry Identifier: Ethics Commitee)
Record Dates: First submitted 2024-03-21; First posted 2024-05-01 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Fibromyalgia; Fatigue; Fatigue; Muscle, Heart; Strength Training; Stress
Keywords: Anxiety; exercise; Strength training; fibromyalgia; healthy individuals; women; neuroinmunoendocrine system
MeSH Terms: conditions — Fibromyalgia; Fatigue; Anxiety Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strength training group with fibromyalgia diagnosis (Experimental): The sample will be composed of 15 subjects (women), aged between 18 and 70 years. Participants must have been diagnosed with fibromyalgia (FM) and/or chronic fatigue syndrome (CFS) at least three months before the start of the study.
  Study participants must not have any other illness and/or injury at the time of the assessments that would prevent them from performing the activity. Likewise, those following pharmacological treatments or any type of cardiorespiratory disease will be excluded from the research.
  Interventions: Behavioral: FMG (Fibromyalgia group)
- Strength training group in no fibromyalgia women (Active Comparator): The sample will be composed of 15 subjects (women), aged between 45 and 70 years. Participants must have not been diagnosed with fibromyalgia. These participants must be healthy individuals.
  Study participants must not have any other illness and/or injury at the time of the assessments that would prevent them from performing the activity. Likewise, those following pharmacological treatments or any type of cardiorespiratory disease will be excluded from the research.
  Interventions: Behavioral: HG (Healthy group)

INTERVENTIONS:
Behavioral: FMG (Fibromyalgia group) — This intervention will report results of a strength training programme in people with fibromyalgia
  Arms: Strength training group with fibromyalgia diagnosis
Behavioral: HG (Healthy group) — This intervention will report results of a strength training programme in people with no fibromyalgia diagnosis
  Arms: Strength training group in no fibromyalgia women

SUMMARY:
Physical exercise is an effective tool for the prevention of various chronic diseases. Fibromyalgia (FM) is a common chronic pain condition, in which patients may also experience a variety of other symptoms, including sleep disturbances, fatigue, stiffness, frequent episodes of pain and mental health problems, as well as possible gastrointestinal disorders. Furthermore, according to the American College of Rheumatology, such a generalised non-joint pain state occurs for at least three months in duration, predominantly in women over 50 years of age. In turn, chronic fatigue syndrome (CFS) presents as a disease characterised by persistent and debilitating fatigue lasting at least six months.

The origin of FM and CFS is unknown, although alterations in the central nervous system (CNS), as well as abnormalities in muscle physiology and immune/inflammatory response are suggested as the main causes.

In addition, most patients with FM are sedentary and in poor physical condition, exacerbated by pain, fatigue or depression, which can limit their daily activities and affect their quality of life and work opportunities. In this regard, physical exercise is considered the most important non-pharmacological strategy for the treatment of FM; however, many clinically relevant questions remain unanswered regarding the most effective approach to exercise therapy in FM patients.

Therefore, the main objective of this project is to analyse the possible physical and mental benefits of a physical exercise programme in people diagnosed with fibromyalgia and/or chronic fatigue syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Women previously diagnosed with fibromyalgia and healthy women aged 18-75 years.
* Not be undertaking any physical activity or exercise programme for at least three months prior to the start of the protocol.

Exclusion Criteria:

* Participants in the study may not present any other illness and/or injury at the time of the assessments that would prevent them from carrying out the activity. In the same way, those following pharmacological treatments or any type of cardiorespiratory disease will be excluded from the research.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
PRE-TEST Time up and go test (TUG test) | 7 days before protocol starts
  The test volunteers will be seated upright in a chair that could be adjusted to suit their leg length, with their legs bent at a 90-degree angle and their arms folded across their chests. Participants were to get up from their seats, move three meters forward, turn around, walk back to the starting point, and then sit down again. Using video capturing, the fastest time between the two trials was found and utilized for analysis
PRE-TEST 5 Times Sit to stand test (5TSTS) | 7 days before protocol starts
  The 5-times sit-to-stand test assesses the lower limb strength, transitional movements, balance and physical performance of older people. Test subjects were positioned upright in a chair that could be adjusted according to the length of their lower limbs, with their arms crossed over their chests and their legs bent to a 90-degree angle. Participants had to perform a total of five full squats in which the total execution time will be recorded.
PRE TEST 10 meters walk test | 7 days before protocol starts
  Participants will be instructed to walk 10 m (marked by taped lines) as quickly as possible without running. The test will be repeated after 2 minutes of rest. Verbal encouragement will be given throughout the test. Two photocells (Witty, Microgate, Italy) will be placed at 6 and 10 m to record the walking time. The shortest running time will be used for analysis
PRE TEST 2 minutes walk | 7 days before protocol starts
  Participants will walk for 2 minutes at the maximum speed they can sustain during that time. The test takes place on a rectangular track (40 x 20 m) with the corners defined by cones. Subjects will be allowed to rest if they need to, but time will not be stopped during their rest period. The total distance (m) covered after 6 min of walking will be measured. All participants will be accompanied by the investigator during the test, but will not be allowed to engage in conversation.
PRE TEST Upper body dinamometry | 7 days before protocol starts
  The dynamometer TKK 5105 (Takei Scientific Instruments Co., Ltd., Niigata, Japan) will be a typical analog handgrip dynamometer with an adjustable handle. This dynamometer will be used to assess the strength of the handgrip. The participant will be placed in a standing position, with the arms parallel but not touching the body, the shoulder adducted and neutrally rotated, and handgrip strength will be measured. The gadget handle will be modified to fit the size of the participants' hands so that each hand's index finger will be 90 degrees bent from the proximal to middle phalangeal joint. Every side will undergo two trials, alternately, with at least a minute of rest in between each session.
PRE TEST Lower body dinamometry | 7 days before protocol starts
  Participants will be seated on the isokinetic dynamometer chair (Biodex Medical System, NY) with both legs flexed at 90° and the testing leg's ankle will be strapped directly to a customized apparatus with a load cell (Model SML500, Interface Scottsdale, AZ, USA). To warm up, each subject will perform 3 progressive MVICs with 3 min of rest between attempts. To assess RFD in each leg, verbal encouragement will be given to the participants to apply "as much force as possible, as fast as possible" throughout the 2 consecutive maximal contractions. RFD will be analyzed using the time interval 0-200 (RFDlate). Subsequently, participants will perform 2 MVICs, each lasting for 5 s with 3 min of rest between contractions, with verbal encouragement. Maximal torque (MVIC) and time to peak voluntary torque (time-to-MVIC) will be evaluated. The right leg will always be evaluated first, and the trial with the highest value will be used for both RFD and MVIC.
PRE TEST Sleep assessment: Karolinska Sleepiness Diary | 7 days before protocol starts
  The Karolinska Sleepiness Diary (KSD) will measure subjective sleep quality (Akerstedt et al., 1994). The KSD will be administered upon awakening in the morning following each of the training sessions (low and high intensity) assessing the following factors using a Likert scale: feeling of rest (1= no rest at all; 3= completely rested); sleep quality (1= very poor; 5= very good); sleep comfort (1= very restless; 5= very calm/relax); ease of falling asleep (1= very difficult; 5= very easy); waking up (1= woken up too early; 3= woken up late); ease of waking up (1= very difficult; 5= very easy); and did you get enough sleep (1= no, definitely very poor; 5= Yes, definitely enough). The higher the score, the higher the quality of sleep will be recorded.
PRE TEST Beck Depression Inventory | 7 days before protocol starts
  Spanish version (Sanz et al., 2003) of the Beck Depression Inventory (BDI) aimed at determining possible signs of depression in the past week. Higher scores indicate higher levels of depression.
PRE TEST State-Trait Anxiety Inventory | 7 days before protocol starts
  State-Trait Anxiety and Trait Anxiety Inventory (STAI), to analyse the levels of anxiety presented at a specific time and in general. Spanish version of Buela-Casal & Guillén-Riquelme (2017). Higher scores indicate higher levels of anxiety.
PRE TEST Perceived stress scale | 7 days before protocol starts
  The Perceived Stress Scale (PSS), to assess the frequency with which participants experience stressful situations and thoughts in the last month. Higher scores indicate higher levels of stress. Remor (2006) was used in its Spanish version.
PRE TEST Pain and fatigue Inventory | 7 days before protocol starts
  -Brief Pain Inventory (BPI). Used to determine the intensity and interference of pain in daily activities. The higher the pain perception, the higher the score obtained. The Spanish version of Badía et al. (2003) was used. -Brief Fatigue Inventory (BFI). This questionnaire measures the intensity of fatigue in the last 24 hours and its interference with daily activities and work. The higher the perception of fatigue, the higher the score obtained (Valenzuela et al., 2002).
PRE TEST Pittsburgh Sleep Quality Questionnaire (PSQI) | 7 days before protocol starts
  Pittsburgh Sleep Quality Questionnaire (PSQI). This questionnaire analyses various parameters related to subjective sleep quality: latency, duration, efficiency and disturbances, as well as consumption of sleeping pills. The Spanish version of the PSQI was used, Hita-Contreras et al.
PRE TEST FIQ (Fibromyalgia Impact Questionnaire) | 7 days before protocol starts
  FIQ (Fibromyalgia Impact Questionnaire). The Spanish version of Rivera & González (2004) was used to assess the impact of fibromyalgia on physical and mental functions (pain, tiredness, fatigue, stiffness, anxiety and depression). Higher scores indicate a worse health condition.
PRE TEST Ergospirometry | 7 days before protocol starts
  The incremental protocol will include a 3-minute warm-up (4.5 km-h -1) followed by an increase to 6 km-h -1, with 1 km-h -1 increments every 45 seconds until exhaustion. Heart rate and the different spirometric variables, including respiratory exchange ratio (RER) and V̇O2 will be constantly monitored. The breath-by-breath method will be used to collect ventilation data during the incremental exercise test for individual assessment of maximal oxygen consumption capacity. The volume transducer and the Vyntus TM CPX gas analyser (Vyaire medical, INC, Hoechberg, Germany) shall be calibrated according to the manufacturer's instructions prior to each test.
PRE TEST Heart Rate Variability (HRV) | 7 days before protocol starts
  HRV analysis. HRV analysis will be performed using a Polar H7 heart rate sensor (Kempele, Finland) to measure R-R intervals during the night at pre- and post-confinement. Analysis of HRV variables will be performed with Kubios HRV 3.0 software (Kuopio, Finland). Additionally, and if necessary, artefact correction will be performed with the same software by applying very low, low or medium threshold filters.
PRE TEST BLOOD EXTRACTION | 7 days before protocol starts
  To carry out the blood extraction, a qualified person will perform a sterile puncture in the cubitus median vein. After 15 minutes of extraction (in the case of serum, essential to facilitate clot formation), both tubes are centrifuged for 10 minutes at 1,600 rpm and at 22ºC. By this process, serum or plasma is isolated in the corresponding tubes and then aliquoted into eppendorf tubes with a total volume of 400 μl in each tube. The serum and plasma samples must be gradually frozen as they are obtained, until they are finally stored at -80ºC.
PRE TEST Balance test | 7 days before protocol starts
  Determination of monopodal and bipodal equilibrium levels.
POST-TEST Time up and go test (TUG test) | 7 days after protocol ends
  The test volunteers will be seated upright in a chair that could be adjusted to suit their leg length, with their legs bent at a 90-degree angle and their arms folded across their chests. Participants were to get up from their seats, move three meters forward, turn around, walk back to the starting point, and then sit down again. Using video capturing, the fastest time between the two trials was found and utilized for analysis
POST-TEST 5 Times Sit to stand test (5TSTS) | 7 days after protocol ends
  The 5-times sit-to-stand test assesses the lower limb strength, transitional movements, balance and physical performance of older people. Test subjects were positioned upright in a chair that could be adjusted according to the length of their lower limbs, with their arms crossed over their chests and their legs bent to a 90-degree angle. Participants had to perform a total of five full squats in which the total execution time will be recorded.
POST TEST 10 meters walk test | 7 days after protocol ends
  Participants will be instructed to walk 10 m (marked by taped lines) as quickly as possible without running. The test will be repeated after 2 minutes of rest. Verbal encouragement will be given throughout the test. Two photocells (Witty, Microgate, Italy) will be placed at 6 and 10 m to record the walking time. The shortest running time will be used for analysis
POST TEST 2 minutes walk | 7 days after protocol ends
  Participants will walk for 2 minutes at the maximum speed they can sustain during that time. The test takes place on a rectangular track (40 x 20 m) with the corners defined by cones. Subjects will be allowed to rest if they need to, but time will not be stopped during their rest period. The total distance (m) covered after 6 min of walking will be measured. All participants will be accompanied by the investigator during the test, but will not be allowed to engage in conversation.
POST TEST Upper body dinamometry | 7 days after protocol ends
  The dynamometer TKK 5105 (Takei Scientific Instruments Co., Ltd., Niigata, Japan) will be a typical analog handgrip dynamometer with an adjustable handle. This dynamometer will be used to assess the strength of the handgrip. The participant will be placed in a standing position, with the arms parallel but not touching the body, the shoulder adducted and neutrally rotated, and handgrip strength will be measured. The gadget handle will be modified to fit the size of the participants' hands so that each hand's index finger will be 90 degrees bent from the proximal to middle phalangeal joint. Every side will undergo two trials, alternately, with at least a minute of rest in between each session.
POST TEST Lower body dinamometry | 7 days after protocol ends
  Participants will be seated on the isokinetic dynamometer chair (Biodex Medical System, NY) with both legs flexed at 90° and the testing leg's ankle will be strapped directly to a customized apparatus with a load cell (Model SML500, Interface Scottsdale, AZ, USA). To warm up, each subject will perform 3 progressive MVICs with 3 min of rest between attempts. To assess RFD in each leg, verbal encouragement will be given to the participants to apply "as much force as possible, as fast as possible" throughout the 2 consecutive maximal contractions. RFD will be analyzed using the time interval 0-200 (RFDlate). Subsequently, participants will perform 2 MVICs, each lasting for 5 s with 3 min of rest between contractions, with verbal encouragement. Maximal torque (MVIC) and time to peak voluntary torque (time-to-MVIC) will be evaluated. The right leg will always be evaluated first, and the trial with the highest value will be used for both RFD and MVIC.
POST TEST Sleep assessment: Karolinska Sleepiness Diary | 7 days after protocol ends
  The Karolinska Sleepiness Diary (KSD) will measure subjective sleep quality (Akerstedt et al., 1994). The KSD will be administered upon awakening in the morning following each of the training sessions (low and high intensity) assessing the following factors using a Likert scale: feeling of rest (1= no rest at all; 3= completely rested); sleep quality (1= very poor; 5= very good); sleep comfort (1= very restless; 5= very calm/relax); ease of falling asleep (1= very difficult; 5= very easy); waking up (1= woken up too early; 3= woken up late); ease of waking up (1= very difficult; 5= very easy); and did you get enough sleep (1= no, definitely very poor; 5= Yes, definitely enough). The higher the score, the higher the quality of sleep will be recorded.
POST TEST Beck Depression Inventory | 7 days after protocol ends
  Spanish version (Sanz et al., 2003) of the Beck Depression Inventory (BDI) aimed at determining possible signs of depression in the past week. Higher scores indicate higher levels of depression.
POST TEST State-Trait Anxiety Inventory | 7 days after protocol ends
  State-Trait Anxiety and Trait Anxiety Inventory (STAI), to analyse the levels of anxiety presented at a specific time and in general. Spanish version of Buela-Casal & Guillén-Riquelme (2017). Higher scores indicate higher levels of anxiety.
POST TEST Perceived stress scale | 7 days after protocol ends
  The Perceived Stress Scale (PSS), to assess the frequency with which participants experience stressful situations and thoughts in the last month. Higher scores indicate higher levels of stress. Remor (2006) was used in its Spanish version.
POST TEST Pain and fatigue Inventory | 7 days after protocol ends
  -Brief Pain Inventory (BPI). Used to determine the intensity and interference of pain in daily activities. The higher the pain perception, the higher the score obtained. The Spanish version of Badía et al. (2003) was used. -Brief Fatigue Inventory (BFI). This questionnaire measures the intensity of fatigue in the last 24 hours and its interference with daily activities and work. The higher the perception of fatigue, the higher the score obtained (Valenzuela et al., 2002).
POST TEST Pittsburgh Sleep Quality Questionnaire (PSQI) | 7 days after protocol ends
  Pittsburgh Sleep Quality Questionnaire (PSQI). This questionnaire analyses various parameters related to subjective sleep quality: latency, duration, efficiency and disturbances, as well as consumption of sleeping pills. The Spanish version of the PSQI was used, Hita-Contreras et al.
POST TEST FIQ (Fibromyalgia Impact Questionnaire) | 7 days after protocol ends
  FIQ (Fibromyalgia Impact Questionnaire). The Spanish version of Rivera & González (2004) was used to assess the impact of fibromyalgia on physical and mental functions (pain, tiredness, fatigue, stiffness, anxiety and depression). Higher scores indicate a worse health condition.
POST TEST Ergospirometry | 7 days after protocol ends
  The incremental protocol will include a 3-minute warm-up (4.5 km-h -1) followed by an increase to 6 km-h -1, with 1 km-h -1 increments every 45 seconds until exhaustion. Heart rate and the different spirometric variables, including respiratory exchange ratio (RER) and V̇O2 will be constantly monitored. The breath-by-breath method will be used to collect ventilation data during the incremental exercise test for individual assessment of maximal oxygen consumption capacity. The volume transducer and the Vyntus TM CPX gas analyser (Vyaire medical, INC, Hoechberg, Germany) shall be calibrated according to the manufacturer's instructions prior to each test.
POST TEST Heart Rate Variability (HRV) | 7 days after protocol ends
  HRV analysis. HRV analysis will be performed using a Polar H7 heart rate sensor (Kempele, Finland) to measure R-R intervals during the night at pre- and post-confinement. Analysis of HRV variables will be performed with Kubios HRV 3.0 software (Kuopio, Finland). Additionally, and if necessary, artefact correction will be performed with the same software by applying very low, low or medium threshold filters.
POST TEST BLOOD EXTRACTION | 7 days after protocol ends
  To carry out the blood extraction, a qualified person will perform a sterile puncture in the cubitus median vein. After 15 minutes of extraction (in the case of serum, essential to facilitate clot formation), both tubes are centrifuged for 10 minutes at 1,600 rpm and at 22ºC. By this process, serum or plasma is isolated in the corresponding tubes and then aliquoted into eppendorf tubes with a total volume of 400 μl in each tube. The serum and plasma samples must be gradually frozen as they are obtained, until they are finally stored at -80ºC.
POST TEST Balance test | 7 days after protocol ends
  Determination of monopodal and bipodal equilibrium levels.

SECONDARY OUTCOMES:
ACUTE PRE-TEST Time up and go test (TUG test) | 5 week since the start of the protocol
  The test volunteers will be seated upright in a chair that could be adjusted to suit their leg length, with their legs bent at a 90-degree angle and their arms folded across their chests. Participants were to get up from their seats, move three meters forward, turn around, walk back to the starting point, and then sit down again. Using video capturing, the fastest time between the two trials was found and utilized for analysis
ACUTE POST-TEST Time up and go test (TUG test) | 5 week since the start of the protocol
  The test volunteers will be seated upright in a chair that could be adjusted to suit their leg length, with their legs bent at a 90-degree angle and their arms folded across their chests. Participants were to get up from their seats, move three meters forward, turn around, walk back to the starting point, and then sit down again. Using video capturing, the fastest time between the two trials was found and utilized for analysis
ACUTE PRE-TEST 5 Times Sit to stand test (5TSTS) | 5 week since the start of the protocol
  The 5-times sit-to-stand test assesses the lower limb strength, transitional movements, balance and physical performance of older people. Test subjects were positioned upright in a chair that could be adjusted according to the length of their lower limbs, with their arms crossed over their chests and their legs bent to a 90-degree angle. Participants had to perform a total of five full squats in which the total execution time will be recorded.
ACUTE POST-TEST 5 Times Sit to stand test (5TSTS) | 5 week since the start of the protocol
  The 5-times sit-to-stand test assesses the lower limb strength, transitional movements, balance and physical performance of older people. Test subjects were positioned upright in a chair that could be adjusted according to the length of their lower limbs, with their arms crossed over their chests and their legs bent to a 90-degree angle. Participants had to perform a total of five full squats in which the total execution time will be recorded.
ACUTE PRE TEST 10 meters walk test | 5 week since the start of the protocol
  Participants will be instructed to walk 10 m (marked by taped lines) as quickly as possible without running. The test will be repeated after 2 minutes of rest. Verbal encouragement will be given throughout the test. Two photocells (Witty, Microgate, Italy) will be placed at 6 and 10 m to record the walking time. The shortest running time will be used for analysis
ACUTE POST TEST 10 meters walk test | 5 week since the start of the protocol
  Participants will be instructed to walk 10 m (marked by taped lines) as quickly as possible without running. The test will be repeated after 2 minutes of rest. Verbal encouragement will be given throughout the test. Two photocells (Witty, Microgate, Italy) will be placed at 6 and 10 m to record the walking time. The shortest running time will be used for analysis
ACUTE PRE TEST Upper body dinamometry | 5 week since the start of the protocol
  The dynamometer TKK 5105 (Takei Scientific Instruments Co., Ltd., Niigata, Japan) will be a typical analog handgrip dynamometer with an adjustable handle. This dynamometer will be used to assess the strength of the handgrip. The participant will be placed in a standing position, with the arms parallel but not touching the body, the shoulder adducted and neutrally rotated, and handgrip strength will be measured. The gadget handle will be modified to fit the size of the participants' hands so that each hand's index finger will be 90 degrees bent from the proximal to middle phalangeal joint. Every side will undergo two trials, alternately, with at least a minute of rest in between each session.
ACUTE POST TEST Upper body dinamometry | 5 week since the start of the protocol
  The dynamometer TKK 5105 (Takei Scientific Instruments Co., Ltd., Niigata, Japan) will be a typical analog handgrip dynamometer with an adjustable handle. This dynamometer will be used to assess the strength of the handgrip. The participant will be placed in a standing position, with the arms parallel but not touching the body, the shoulder adducted and neutrally rotated, and handgrip strength will be measured. The gadget handle will be modified to fit the size of the participants' hands so that each hand's index finger will be 90 degrees bent from the proximal to middle phalangeal joint. Every side will undergo two trials, alternately, with at least a minute of rest in between each session.
ACUTE PRE TEST Lower body dinamometry | 5 week since the start of the protocol
  Participants will be seated on the isokinetic dynamometer chair (Biodex Medical System, NY) with both legs flexed at 90° and the testing leg's ankle will be strapped directly to a customized apparatus with a load cell (Model SML500, Interface Scottsdale, AZ, USA). To warm up, each subject will perform 3 progressive MVICs with 3 min of rest between attempts. To assess RFD in each leg, verbal encouragement will be given to the participants to apply "as much force as possible, as fast as possible" throughout the 2 consecutive maximal contractions. RFD will be analyzed using the time interval 0-200 (RFDlate). Subsequently, participants will perform 2 MVICs, each lasting for 5 s with 3 min of rest between contractions, with verbal encouragement. Maximal torque (MVIC) and time to peak voluntary torque (time-to-MVIC) will be evaluated. The right leg will always be evaluated first, and the trial with the highest value will be used for both RFD and MVIC.
ACUTE POST TEST Lower body dinamometry | 5 week since the start of the protocol
  Participants will be seated on the isokinetic dynamometer chair (Biodex Medical System, NY) with both legs flexed at 90° and the testing leg's ankle will be strapped directly to a customized apparatus with a load cell (Model SML500, Interface Scottsdale, AZ, USA). To warm up, each subject will perform 3 progressive MVICs with 3 min of rest between attempts. To assess RFD in each leg, verbal encouragement will be given to the participants to apply "as much force as possible, as fast as possible" throughout the 2 consecutive maximal contractions. RFD will be analyzed using the time interval 0-200 (RFDlate). Subsequently, participants will perform 2 MVICs, each lasting for 5 s with 3 min of rest between contractions, with verbal encouragement. Maximal torque (MVIC) and time to peak voluntary torque (time-to-MVIC) will be evaluated. The right leg will always be evaluated first, and the trial with the highest value will be used for both RFD and MVIC.
ACUTE PRE TEST Sleep assessment: Karolinska Sleepiness Diary | 5 week since the start of the protocol
  The Karolinska Sleepiness Diary (KSD) will measure subjective sleep quality (Akerstedt et al., 1994). The KSD will be administered upon awakening in the morning following each of the training sessions (low and high intensity) assessing the following factors using a Likert scale: feeling of rest (1= no rest at all; 3= completely rested); sleep quality (1= very poor; 5= very good); sleep comfort (1= very restless; 5= very calm/relax); ease of falling asleep (1= very difficult; 5= very easy); waking up (1= woken up too early; 3= woken up late); ease of waking up (1= very difficult; 5= very easy); and did you get enough sleep (1= no, definitely very poor; 5= Yes, definitely enough). The higher the score, the higher the quality of sleep will be recorded.
ACUTE POST TEST Sleep assessment: Karolinska Sleepiness Diary | 5 week since the start of the protocol
  The Karolinska Sleepiness Diary (KSD) will measure subjective sleep quality (Akerstedt et al., 1994). The KSD will be administered upon awakening in the morning following each of the training sessions (low and high intensity) assessing the following factors using a Likert scale: feeling of rest (1= no rest at all; 3= completely rested); sleep quality (1= very poor; 5= very good); sleep comfort (1= very restless; 5= very calm/relax); ease of falling asleep (1= very difficult; 5= very easy); waking up (1= woken up too early; 3= woken up late); ease of waking up (1= very difficult; 5= very easy); and did you get enough sleep (1= no, definitely very poor; 5= Yes, definitely enough). The higher the score, the higher the quality of sleep will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad Deporte Universidad Católica San Antonio de Murcia, Murcia, España, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The data will be available upon request via email to the principal investigator, in this case Carmen Daniela Quero (cdquero@ucam.edu).